CLINICAL TRIAL: NCT02137707
Title: An Investigator-initiated, Multicenter, Phase IV, Open-label Study to Evaluate the Biological Basis for Disease Progression in Relapsing-remitting Multiple Sclerosis Patients Treated in Routine Practice With Gilenya for 2 Years
Brief Title: Biologic Basis for Multiple Sclerosis Disease Progression in RRMS Patients Treated With Gilenya
Acronym: IGLOO
Status: Completed | Type: Observational
Sponsor: McGill University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Jack Antel, Professor, M.D., McGill University
Other Study IDs: CFTY720DCA04T
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Multiple Sclerosis-Relapsing-Remitting
Keywords: Multiple Sclerosis, Relapsing-Remitting; Gilenya; Fingolimod
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, peripheral blood mononuclear cells, DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gilenya treatment: Gilenya oral form once a day
  Interventions: Drug: Gilenya

INTERVENTIONS:
Drug: Gilenya — All patients will receive Gilenya
  Other Names: fingolimod

SUMMARY:
This study will determine whether in RRMS patients receiving Gilenya there is a link between disease progression and biologic markers.

DETAILED DESCRIPTION:
The biologic basis that determines disease progression in multiple sclerosis (MS) patients remains to be defined. We propose that a long term study of patients where inflammatory activity of the disease is expected to be controlled on treatment, will identify patients into cohorts of those whose disease is deemed to be stable with those patients whose disease has been deemed to progress. Once the two groups have been identified, it will then be possible to assess whether there are differences in biologic markers between the two groups. These markers would then have the potential to be used to monitor disease progression or be predictors for patient response to drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Deemed by the subject's treating physician to be a suitable candidate for Gilenya therapy in accordance with the Canadian Product Monograph for Gilenya
* has an overall EDSS not above 7.0
* is not currently receiving Gilenya
* is able to perform adequately for EDSS assessment and cognitive tests
* is able to undergo a MRI
* is able to provide blood samples

Exclusion Criteria:

* is over 65 years of age and under 18 years of age
* has less than 4 weeks of discontinuation with steroid treatment for a relapse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsing-remitting multiple sclerosis deemed by their treating physician to be a suitable candidate for Gilenya therapy
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2012-11; Primary Completion 2017-11 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Determination of disease progression of subjects treated with Gilenya over 2 years | 2 years
  Changes in number of new and enlarging T2 lesions by MRI between baseline and Year 2 will be compared with immune biomarkers (Teff:Treg ratio)

SECONDARY OUTCOMES:
Change in cognitive function in patients treated with Gilenya | 2 years
  changes in brain volume assessed by MRI between baseline and Year 2 will be compared with immune biomarkers
Changes in biologic measures in patients treated with Gilenya | 2 years
  change in MTR MRI as assessment of myelin content will be compared with blood biomarkers
Safety and tolerability of Gilenya therapy will be assessed | 2 years
  Safety parameters include the initial cardiac effects, liver function, infections and migraines/headaches

CONTACTS AND LOCATIONS:
Overall Officials: Jack Antel, MD, Principal Investigator — McGill University; Amit Bar-Or, MD, Principal Investigator — McGill University
Locations (6):
- Canada (6):
  - University of British Columbia, Vancouver, British Columbia
  - Dalhousie University Multiple Sclerosis Research Unit, Halifax, Nova Scotia
  - Ottawa General Hospital, Ottawa, Ontario
  - Clinique Neuro Rive-Sud, Greenfield Park, Quebec
  - Montreal Neurological Institute, Montreal, Quebec
  - Centre hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec

REFERENCES:
- [Derived] Ghadiri M, Rezk A, Li R, Evans A, Giacomini PS, Barnett MH, Antel J, Bar-Or A. Pre-treatment T-cell subsets associate with fingolimod treatment responsiveness in multiple sclerosis. Sci Rep. 2020 Jan 15;10(1):356. doi: 10.1038/s41598-019-57114-2. PMID 31941953